CLINICAL TRIAL: NCT02378753
Title: [rVSVΔG-ZEBOV] Ebola Prevention Vaccine Evaluation in Sierra Leone
Brief Title: STRIVE (Sierra Leone Trial to Introduce a Vaccine Against Ebola)
Acronym: STRIVE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Sierra Leone (Other); Ministry of Health and Sanitation, Sierra Leone (Other Government); Department of Health and Human Services (U.S. Federal Agency); eHealth Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCIRD-6689
Record Dates: First submitted 2015-02-19; First posted 2015-03-04 (Estimated); Results first posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2016-07

CONDITIONS: Hemorrhagic Fever, Ebola
Keywords: Ebola; Sierra Leone; vaccine; rVSVΔG-ZEBOV
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- rVSVΔG-ZEBOV (immediate vaccination) (Experimental): One intramuscular (deltoid) injection of rVSVΔG-ZEBOV (2 x 10^7 plaque forming units)
  Interventions: Biological: rVSVΔG-ZEBOV
- rVSVΔG-ZEBOV (deferred vaccination) (Experimental): One intramuscular (deltoid) injection of rVSVΔG-ZEBOV (2 x 10^7 plaque forming units) in participants randomized to receive deferred vaccination (18-24 weeks after enrollment).
  Interventions: Biological: rVSVΔG-ZEBOV

INTERVENTIONS:
Biological: rVSVΔG-ZEBOV — The rVSVΔG-ZEBOV vaccine is comprised of a single recombinant VSV isolate (11481 nontypeable) modified to replace the gene encoding the G envelope GP with the gene encoding the envelope GP from ZEBOV (Kikwit, 1995 strain).
  Other Names: BPSC-1001

SUMMARY:
The 2014 outbreak of Ebola in West Africa is the largest in recorded history with widespread and intense transmission in Guinea, Liberia, and Sierra Leone. The high infectivity of blood and secretions, lack of appropriate personal protective equipment (PPE) and challenges in following infection control and prevention protocols put healthcare workers at high risk during outbreaks, and direct contact with the bodies of deceased Ebola victims can also sustain community transmission. This study will accelerate introduction and use of monovalent recombinant vesicular stomatitis virus Ebola vaccine (rVSVΔG-ZEBOV) among healthcare workers and frontline personnel involved in the Ebola outbreak response in Sierra Leone, while concurrently evaluating the safety and efficacy of the vaccine.

This is an unblinded, randomized trial with phased vaccine introduction in the target population. Participation in the study will be voluntary and open to adults 18 years of age and older who are at high risk of exposure to Ebola infection through their daily work and who work in a selected study area.

DETAILED DESCRIPTION:
The Ebola outbreak was confirmed in March 2014 with widespread and intense transmission in Guinea, Liberia, and Sierra Leone. While there are no U.S. Food and Drug Administration (FDA)-approved pharmaceuticals to prevent or treat Ebola, two candidate vaccines are being tested in humans for dosing, tolerability, and safety. This study will evaluate monovalent recombinant vesicular stomatitis virus Ebola vaccine that remains replication competent (rVSVΔG-ZEBOV) in Sierra Leone.

The high infectivity of blood and secretions, lack of appropriate personal protective equipment (PPE) and challenges in following infection control and prevention protocols put healthcare workers at high risk during outbreaks, and direct contact with the bodies of deceased Ebola victims can also sustain community transmission.

This unblinded, randomized trial will evaluate vaccine efficacy (VE) and safety with phased vaccine introduction in the target population. Participation in the study will be voluntary and open to adults 18 years of age and older who are at high risk of exposure to Ebola infection through their daily work and who work in a selected study area. This includes: 1) personnel working in healthcare facilities where care is provided for Ebola patients; 2) personnel working in non-Ebola healthcare facilities who may have exposure to undiagnosed Ebola-infected individuals; and 3) personnel working in one of the following job categories: surveillance team, ambulance team, or laboratory worker responsible for swabbing deceased persons. Staff members involved in this study are also eligible to receive the vaccine under this protocol; study staff will be followed for 6 months post-vaccination to monitor for safety of rVSVΔG-ZEBOV.

Eligible participants within a healthcare facility or frontline team will be enrolled and individually randomized to either immediate or deferred vaccination. A single dose of rVSVΔG-ZEBOV will be administered intramuscularly. Immediate vaccination is defined as vaccination within 7 days of enrollment and deferred vaccination is defined as vaccination at the end of an 18-24 week follow-up period. Participants will not be blinded to the randomized assignment of immediate or deferred vaccination. All enrolled participants will have the opportunity to receive rVSVΔG-ZEBOV by the end of the study. Enrollment and vaccination will be phased over time.

Ebola events that occur during the 18-24 week post-enrollment will be included in the VE analysis, with the immediate vaccination arm contributing vaccinated follow-up time and the deferred vaccination arm contributing unvaccinated follow-up time. All participants, regardless of randomized assignment, will be followed for 6 months after vaccination to monitor for safety of rVSVΔG-ZEBOV.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Member of target population at the time of enrollment:

   * active worker in an Ebola care, holding, or treatment center (may include physicians, nurses, nurse aides, lab technicians, pharmacists, pharmacy technicians, cleaners, and security and administrative staff);
   * active worker in a facility providing non-Ebola-related healthcare (may include physicians, nurses, nurse aides, lab technicians, pharmacists, pharmacy technicians, cleaners, and security and administrative staff);
   * active frontline worker in one of the following job categories: surveillance team, ambulance team, burial worker, or worker responsible for swabbing deceased persons.
3. Reasonably anticipates living in Sierra Leone for the 18-24 weeks following enrollment.
4. Reachable by phone throughout the 6 month post-vaccination safety follow-up period.
5. Willing to adhere to personal protective equipment (PPE) and infection control recommendations.
6. Able and willing to complete the informed consent process and study procedures.
7. Willing to receive vaccine in either the immediate or the deferred trial arms, according to random assignment.

Exclusion Criteria:

1. History of Ebola (self-report).
2. Prior receipt of experimental Ebola or Marburg vaccine.
3. History of human immunodeficiency virus (HIV) or clinically important immunodeficiency (self-report).
4. Any history of allergy or anaphylaxis to prior vaccines
5. Breast-feeding an infant or child.
6. Any reason the investigator suspects that data collected from this person would be incomplete or of poor quality.
7. Current pregnancy (a negative urine pregnancy test is required for women participants <50 years of age who self-report as not pregnant).
8. Currently being followed for known exposure to Ebola.
9. Known experimental research agents or other vaccine within 28 days (4 weeks) before vaccination.
10. Fever ≥ 38.0°C (100.4°F) at time of vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8651 (Actual)
Dates: Start 2015-04; Primary Completion 2016-11-08 (Actual); Study Completion 2016-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Samai, MBChB,PhD, Principal Investigator — University of Sierra Leone
Locations (5):
- Sierra Leone (5):
  - College of Medicine and Allied Health Sciences (COMAHS), Freetown, Western Area Urban
  - Bombali, Bombali District
  - Port Loko, Port Loko District
  - Tonkolili, Tonkolili District
  - Western Area Rural, Western Area District

REFERENCES:
- [Derived] Simon JK, Kennedy SB, Mahon BE, Dubey SA, Grant-Klein RJ, Liu K, Hartzel J, Coller BG, Welebob C, Hanson ME, Grais RF. Immunogenicity of rVSVDeltaG-ZEBOV-GP Ebola vaccine (ERVEBO(R)) in African clinical trial participants by age, sex, and baseline GP-ELISA titer: A post hoc analysis of three Phase 2/3 trials. Vaccine. 2022 Nov 2;40(46):6599-6606. doi: 10.1016/j.vaccine.2022.09.037. Epub 2022 Oct 5. PMID 36208978
- [Derived] Legardy-Williams JK, Carter RJ, Goldstein ST, Jarrett OD, Szefer E, Fombah AE, Tinker SC, Samai M, Mahon BE. Pregnancy Outcomes among Women Receiving rVSVDelta-ZEBOV-GP Ebola Vaccine during the Sierra Leone Trial to Introduce a Vaccine against Ebola. Emerg Infect Dis. 2020 Mar;26(3):541-548. doi: 10.3201/eid2603.191018. Epub 2020 Mar 17. PMID 32017677
- [Derived] Kabineh AK, Carr W, Motevalli M, Legardy-Williams J, Vincent W, Mahon BE, Samai M. Operationalizing International Regulatory Standards in a Limited-Resource Setting During an Epidemic: The Sierra Leone Trial to Introduce a Vaccine Against Ebola (STRIVE) Experience. J Infect Dis. 2018 May 18;217(suppl_1):S56-S59. doi: 10.1093/infdis/jiy111. PMID 29788349
- [Derived] Carter RJ, Senesi RGB, Dawson P, Gassama I, Kargbo SAS, Petrie CR, Rogers MH, Samai M, Luman ET. Participant Retention in a Randomized Clinical Trial in an Outbreak Setting: Lessons From the Sierra Leone Trial to Introduce a Vaccine Against Ebola (STRIVE). J Infect Dis. 2018 May 18;217(suppl_1):S65-S74. doi: 10.1093/infdis/jiy094. PMID 29788348
- [Derived] Conteh MA, Goldstein ST, Wurie HR, Gidudu J, Lisk DR, Carter RJ, Seward JF, Hampton LM, Wang D, Andersen LE, Arvay M, Schrag SJ, Dawson P, Fombah AE, Petrie CR, Feikin DR, Russell JBW, Lindblad R, Kargbo SAS, Samai M, Mahon BE. Clinical Surveillance and Evaluation of Suspected Ebola Cases in a Vaccine Trial During an Ebola Epidemic: The Sierra Leone Trial to Introduce a Vaccine Against Ebola. J Infect Dis. 2018 May 18;217(suppl_1):S33-S39. doi: 10.1093/infdis/jiy061. PMID 29788347
- [Derived] Jarrett OD, Seward JF, Fombah AE, Lindblad R, Jalloh MI, El-Khorazaty J, Dawson P, Burton D, Zucker J, Carr W, Bah MM, Deen GF, George PM, James F, Lisk DR, Pratt D, Russell JBW, Sandy JD, Turay P, Hamel MJ, Schrag SJ, Walker RE, Samai M, Goldstein ST. Monitoring Serious Adverse Events in the Sierra Leone Trial to Introduce a Vaccine Against Ebola. J Infect Dis. 2018 May 18;217(suppl_1):S24-S32. doi: 10.1093/infdis/jiy042. PMID 29788346
- [Derived] Samai M, Seward JF, Goldstein ST, Mahon BE, Lisk DR, Widdowson MA, Jalloh MI, Schrag SJ, Idriss A, Carter RJ, Dawson P, Kargbo SAS, Leigh B, Bawoh M, Legardy-Williams J, Deen G, Carr W, Callis A, Lindblad R, Russell JBW, Petrie CR, Fombah AE, Kargbo B, McDonald W, Jarrett OD, Walker RE, Gargiullo P, Bash-Taqi D, Gibson L, Fofanah AB, Schuchat A; STRIVE Study Team. The Sierra Leone Trial to Introduce a Vaccine Against Ebola: An Evaluation of rVSV∆G-ZEBOV-GP Vaccine Tolerability and Safety During the West Africa Ebola Outbreak. J Infect Dis. 2018 May 18;217(suppl_1):S6-S15. doi: 10.1093/infdis/jiy020. PMID 29788345
- [Derived] Carter RJ, Idriss A, Widdowson MA, Samai M, Schrag SJ, Legardy-Williams JK, Estivariz CF, Callis A, Carr W, Webber W, Fischer ME, Hadler S, Sahr F, Thompson M, Greby SM, Edem-Hotah J, Momoh RM, McDonald W, Gee JM, Kallon AF, Spencer-Walters D, Bresee JS, Cohn A, Hersey S, Gibson L, Schuchat A, Seward JF. Implementing a Multisite Clinical Trial in the Midst of an Ebola Outbreak: Lessons Learned From the Sierra Leone Trial to Introduce a Vaccine Against Ebola. J Infect Dis. 2018 May 18;217(suppl_1):S16-S23. doi: 10.1093/infdis/jix657. PMID 29788343
- [Derived] Fombah AE, Goldstein ST, Jarrett OD, Jalloh MI, El-Khorazaty J, Lisk DR, Legardy-Williams J, Pratt DA, George PM, Russell JBW, Schrag SJ, Dawson P, Deen GF, Carr W, Lindblad R, James F, Bah MM, Yillia JF, Sandy JD, Turay PE, Conteh MA, Slutsker L, Mahon BE, Samai M, Seward JF. Health Conditions in an Adult Population in Sierra Leone: Data Reported From the Sierra Leone Trial to Introduce a Vaccine Against Ebola (STRIVE). J Infect Dis. 2018 May 18;217(suppl_1):S75-S80. doi: 10.1093/infdis/jix603. PMID 29788342
- [Derived] Callis A, Carter VM, Ramakrishnan A, Albert AP, Conteh L, Barrie AA, Fahnbulleh L, Koroma MM, Saidu S, Williams O, Samai M. Lessons Learned in Clinical Trial Communication During an Ebola Outbreak: The Implementation of STRIVE. J Infect Dis. 2018 May 18;217(suppl_1):S40-S47. doi: 10.1093/infdis/jix558. PMID 29788341
- [Derived] Edem-Hotah J, McDonald W, Abu PM, Luman ET, Carter RJ, Koker A, Goldstein ST. Utilizing Nurses to Staff an Ebola Vaccine Clinical Trial in Sierra Leone during the Ebola Outbreak. J Infect Dis. 2018 May 18;217(suppl_1):S60-S64. doi: 10.1093/infdis/jix389. PMID 29788340
- [Derived] Jusu MO, Glauser G, Seward JF, Bawoh M, Tempel J, Friend M, Littlefield D, Lahai M, Jalloh HM, Sesay AB, Caulker AF, Samai M, Thomas V, Farrell N, Widdowson MA. Rapid Establishment of a Cold Chain Capacity of -60 degrees C or Colder for the STRIVE Ebola Vaccine Trial During the Ebola Outbreak in Sierra Leone. J Infect Dis. 2018 May 18;217(suppl_1):S48-S55. doi: 10.1093/infdis/jix336. PMID 29788339
- [Derived] Coller BG, Blue J, Das R, Dubey S, Finelli L, Gupta S, Helmond F, Grant-Klein RJ, Liu K, Simon J, Troth S, VanRheenen S, Waterbury J, Wivel A, Wolf J, Heppner DG, Kemp T, Nichols R, Monath TP. Clinical development of a recombinant Ebola vaccine in the midst of an unprecedented epidemic. Vaccine. 2017 Aug 16;35(35 Pt A):4465-4469. doi: 10.1016/j.vaccine.2017.05.097. Epub 2017 Jun 21. PMID 28647166

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rVSVΔG-ZEBOV (Immediate Vaccination) | rVSVΔG-ZEBOV (Deferred Vaccination)
Started | 4319 | 4332
Completed | 4101 | 3637
Not Completed | 218 | 695

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were re-assessed for participants on the deferred arm when they presented for vaccination (18-24 weeks after randomization/enrollment). The number on the deferred arm reflects the number of deferred participants who returned for vaccination (e.g. did not drop out during the 18-24 week period).
Groups:
- Total: Total of all reporting groups
Arm/Group | rVSVΔG-ZEBOV (Immediate Vaccination) | rVSVΔG-ZEBOV (Deferred Vaccination) | Total
Number analyzed (Participants) | 4319 | 4332 | 8651
Age, Continuous [Median (Full Range); unit: years] | 30.5 [18.1 to 78.0] | 31.0 [18.0 to 79.5] | 30.7 [18.0 to 79.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1703 | 1704 | 3407
  Male | 2616 | 2628 | 5244
Region of Enrollment [Count of Participants; unit: Participants]
  Sierra Leone | 4183 | 3821 | 8004

OUTCOME MEASURES:

1. Primary Outcome: Laboratory-confirmed Ebola (Study Diagnostics)
Description: Incidence of Ebola confirmed by the STRIVE study laboratory in each treatment group during the Randomized Portion of the trial. For the vaccine efficacy endpoint, all enrolled participants in both arms were followed for 18-24 weeks after enrollment (after which point participants in the deferred cohort received crossover vaccination). Statistical analysis was to proceed as survival analysis (time-to-event/time-to-infection) of cohort follow-up data during this period.
  There were no laboratory-confirmed cases of Ebola among study participants, so therefore no efficacy analyses were performed.
Time Frame: > 21 days following vaccination
Population: The Overall Number of Participants Analyzed for this endpoint is the number of participants with suspected Ebola in each group who provided biological samples to the study laboratory for testing.
Measure: Count of Participants; unit: Participants
Arm/Group | rVSVΔG-ZEBOV (Immediate Vaccination) | rVSVΔG-ZEBOV (Deferred Vaccination)
Number analyzed (Participants) | 24 | 10
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Occurrence of Serious Adverse Events During the 6 Months Following the Vaccination
Description: Number of Participants with Occurrence of SAEs within the 6-month follow-up period following a single dose of rVSVΔG-ZEBOV. Vaccination in the immediate group occurred within 7 days of enrollment if possible, and vaccination in the deferred-vaccination group occurred 18-24 weeks after enrollment.
Time Frame: 6 months following vaccination
Population: The Overall Number of Participants Analyzed for this endpoint is the number of participants in each group who provided any safety/AE data during 6-month (18- to 24-week) follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | rVSVΔG-ZEBOV (Immediate Vaccination) | rVSVΔG-ZEBOV (Deferred Vaccination)
Number analyzed (Participants) | 4261 | 3788
Participants | 54 | 47

3. Secondary Outcome: Death Due to Laboratory-confirmed Ebola
Description: Deaths due to Ebola confirmed by the STRIVE study laboratory in each treatment group during the Randomized Portion of the trial. There were no laboratory-confirmed cases of Ebola among study participants, so therefore no efficacy analyses were performed.
Time Frame: 6 months following vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | rVSVΔG-ZEBOV (Immediate Vaccination) | rVSVΔG-ZEBOV (Deferred Vaccination)
Number analyzed (Participants) | 4261 | 3788
Participants | 0 | 0

4. Secondary Outcome: Ebola Confirmed by Non-study or Study Diagnostics
Description: Incidence of Ebola confirmed by the STRIVE study laboratory or by a non-study laboratory in each treatment group during the Randomized Portion of the trial. For the vaccine efficacy endpoint, all enrolled participants in both arms were followed for 18-24 weeks after enrollment (after which point participants in the deferred cohort received crossover vaccination). Statistical analysis was to proceed as survival analysis (time-to-event/time-to-infection) of cohort follow-up data during this period. There were no laboratory-confirmed cases of Ebola among study participants, so therefore no efficacy analyses were performed.
Time Frame: 6 months following vaccination
Population: The Overall Number of Participants Analyzed for this endpoint is the number of participants with suspected Ebola in each group who provided biological samples for testing, whether to the study laboratory or to a non-study laboratory.
Measure: Count of Participants; unit: Participants
Arm/Group | rVSVΔG-ZEBOV (Immediate Vaccination) | rVSVΔG-ZEBOV (Deferred Vaccination)
Number analyzed (Participants) | 52 | 31
Participants | 0 | 0

5. Secondary Outcome: Suspected, Probable or Laboratory-confirmed Ebola
Description: Incidence of suspected, probable, or laboratory-confirmed Ebola, where "suspected" and "probable" cases are defined by the August 9, 2014 World Health Organization case definition recommendations for use during an Ebola outbreak, and laboratory-confirmed Ebola includes both study laboratory and non-study laboratory diagnostics. An Ebola Screening Form was required to be completed for all participants referred for evaluation of suspected Ebola; the Outcome Measure (Count of Participants) reflects the number of participants in each group for whom an Ebola Screening Form was completed.
Time Frame: 6 months following vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | rVSVΔG-ZEBOV (Immediate Vaccination) | rVSVΔG-ZEBOV (Deferred Vaccination)
Number analyzed (Participants) | 4261 | 3788
Participants | 27 | 17

6. Secondary Outcome: Number of Participants With Occurrence of Solicited Injection-site and Systemic Reactogenicity Signs and Symptoms, Including Fever, on Vaccination Day and During the 7 Days Following the Vaccination or Enrollment.
Description: Solicited symptoms were assessed only in safety sub-study participants (the first 449 participants enrolled at the COMAHS Library site), during the 7 days after vaccination (immediate group) or after enrollment without vaccination (deferred group). Participants were actively solicited for the occurrence of local (injection-site) pain, redness, and swelling and the following systemic reactogenicity symptoms: fever, joint pain, joint swelling, muscle pain, fatigue, feeling unwell, chills, headache, vomiting, nausea, diarrhea, abdominal pain, rash, oral ulcers, and skin vesicles (blisters).
Time Frame: Vaccination day and for 7 days following vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | rVSVΔG-ZEBOV (Immediate Vaccination) | rVSVΔG-ZEBOV (Deferred Vaccination)
Number analyzed (Participants) | 217 | 219
Participants | 202 | 76

7. Secondary Outcome: Number of Participants With Occurrence of Solicited and Unsolicited AEs During the 28 Days Following the Vaccination or Enrollment
Description: Solicited local and systemic reactogenicity symptoms and unsolicited adverse events were assessed in safety sub-study participants (the first 449 participants enrolled at the COMAHS Library site), during the 28 days after vaccination (immediate group) or after enrollment without vaccination (deferred group).
Time Frame: During 28 days following vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | rVSVΔG-ZEBOV (Immediate Vaccination) | rVSVΔG-ZEBOV (Deferred Vaccination)
Number analyzed (Participants) | 217 | 219
Participants
  Solicited AEs | 203 | 117
  Unsolicited AEs | 101 | 27

ADVERSE EVENTS:
Time Frame: 6 months after vaccination
Description: Number of Participants with occurrence of SAEs within the 6-month follow-up period following a single dose of rVSVΔG-ZEBOV. Vaccination in the immediate group occurred within 7 days of enrollment if possible, and vaccination in the deferred-vaccination group occurred 18-24 weeks after enrollment. The overall number of participants analyzed is the number of participants in each group who provided any safety/AE data during 6-month (18- to 24-week) follow-up.
Arm/Group | rVSVΔG-ZEBOV (Immediate Vaccination) | rVSVΔG-ZEBOV (Deferred Vaccination)
All-Cause Mortality (participants affected / at risk) | 8/4261 | 11/3788
Serious Adverse Events (participants affected / at risk) | 54/4261 | 47/3788
Other Adverse Events (participants affected / at risk) | 2537/4261 | 1512/3788
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rVSVΔG-ZEBOV (Immediate Vaccination) (N=4261) | rVSVΔG-ZEBOV (Deferred Vaccination) (N=3788)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 3 | 4
Inguinal hernia, obstructive (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 3 | 3
Toothache (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 0 | 1
Drowning (General disorders) | 0 | 1
Electrocution (General disorders) | 1 | 0
Hernia (General disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 1 | 2
Encephalitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 3
HIV wasting syndrome (Infections and infestations) | 1 | 0
Ludwig angina (Infections and infestations) | 1 | 1
Malaria (Infections and infestations) | 12 | 3
Pelvic inflammatory disease (Infections and infestations) | 1 | 2
Pyonephrosis (Infections and infestations) | 0 | 1
Salpingo-oophoritis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Typhoid fever (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Aphasia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Conversion disorder (Psychiatric disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Adnexal torsion (Reproductive system and breast disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
Pelvic adhesions (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rVSVΔG-ZEBOV (Immediate Vaccination) (N=4261) | rVSVΔG-ZEBOV (Deferred Vaccination) (N=3788)
Abdominal pain (Gastrointestinal disorders) | 240 | 200
Asthenia (General disorders) | 361 | 242
Fatigue (General disorders) | 238 | 52
Feeling hot (General disorders) | 403 | 281
Pain (General disorders) | 663 | 370
Pyrexia (General disorders) | 467 | 222
Nasopharyngitis (Infections and infestations) | 232 | 110
Decreased appetite (Metabolism and nutrition disorders) | 354 | 195
Arthralgia (Musculoskeletal and connective tissue disorders) | 530 | 370
Headache (Nervous system disorders) | 1402 | 770
Pruritus (Skin and subcutaneous tissue disorders) | 256 | 138
Rash (Gastrointestinal disorders) | 274 | 155

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No